CLINICAL TRIAL: NCT00023816
Title: Third Phase I and Pharmacokinetic Study Of FB-642 Administered Orally To Patients With Advanced Solid Tumors
Brief Title: Carbendazim in Treating Patients With Advanced Solid Tumors or Lymphoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068867; UCLA-0002007; ILEX-FB-642-103-A4; NCI-G01-2006
Record Dates: First submitted 2001-09-13; First posted 2004-04-05 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2001-12

CONDITIONS: Lymphoma; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: stage IV adult Hodgkin lymphoma; recurrent adult Hodgkin lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; unspecified adult solid tumor, protocol specific; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult Burkitt lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; stage IV adult T-cell leukemia/lymphoma; recurrent adult T-cell leukemia/lymphoma; primary central nervous system non-Hodgkin lymphoma; AIDS-related peripheral/systemic lymphoma; AIDS-related primary CNS lymphoma; intraocular lymphoma; stage IV mantle cell lymphoma; recurrent mantle cell lymphoma; anaplastic large cell lymphoma; stage IV mycosis fungoides/Sezary syndrome; recurrent mycosis fungoides/Sezary syndrome; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Lymphoma; Hodgkin Disease; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Intraocular Lymphoma; Lymphoma, Mantle-Cell; Lymphoma, Large-Cell, Anaplastic; Mycosis Fungoides; Sezary Syndrome; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — carbendazim

INTERVENTIONS:
Drug: carbendazim

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die.

PURPOSE: Phase I trial to study the effectiveness of carbendazim in treating patients who have advanced solid tumors or lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose of carbendazim in patients with advanced solid tumors or lymphoma. II. Determine the qualitative and quantitative toxic effects of this drug in these patients. III. Determine the pharmacokinetics of this drug in these patients. IV. Determine the recommended phase II dose of this drug. V. Determine any antitumor effects of this drug in these patients.

OUTLINE: This is a dose-escalation, multicenter study. Patients receive oral carbendazim 2-3 times daily 5 days a week for 3-4 weeks. Treatment repeats every 4 weeks in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of carbendazim until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Patients are followed at 30 days.

PROJECTED ACCRUAL: Approximately 30-60 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed advanced solid tumor for which no standard therapy exists or which has progressed or recurred after prior therapy OR Lymphoma for which no further therapeutic options exist No hematological malignancies (e.g., leukemia) No known brain or leptomeningeal disease unless previously treated with radiotherapy, not currently treated with corticosteroid therapy, and no clinical symptoms present

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: At least 12 weeks Hematopoietic: Absolute neutrophil count at least 1,000/mm3 Hemoglobin at least 9 g/dL Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 2 mg/dL AST or ALT no greater than 3 times upper limit of normal (ULN) (5 times ULN if due to tumor involvement) Alkaline phosphatase less than 2.5 times ULN Renal: Creatinine no greater than 2 mg/dL OR Creatinine clearance at least 60 mL/min Cardiovascular: No unstable atrial or ventricular arrhythmias that require control by medication No ischemic event within the past 6 months Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception Abnormalities that would affect absorption of study drug allowed at investigator's discretion No other severe disease or psychiatric disorder that would preclude study No phenylketonuria No known hypersensitivity reaction to artificial sweetener aspartame (e.g., Nutrasweet)

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: Recovered from prior chemotherapy for cancer No other concurrent cytotoxic therapy Endocrine therapy: See Disease Characteristics Radiotherapy: See Disease Characteristics Recovered from prior radiotherapy for cancer Surgery: Recovered from prior surgery for cancer Prior gastrointestinal surgery allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Lee S. Rosen, MD, Study Chair — Jonsson Comprehensive Cancer Center